CLINICAL TRIAL: NCT03813082
Title: Age-related Changes in Sleep-wake Regulation: Effects of Sleep Loss on Possible Molecular Markers of Sleep Need
Brief Title: Age-related Changes in Sleep-wake Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PSS-Sleep
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Sleep Deprivation
Keywords: Positron emission tomography; Magnetic resonance spectroscopy; Aging
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep deprivation young men (Experimental): Young study participants will complete four nights in the sleep laboratory, whereas they will stay awake during one night. PET brain imaging will be conducted at the same circadian time on three consecutive afternoons (prior, during and after prolonged wakefulness). Additionally, validated tests of vigilance and cognitive performance will be administered and the brain waves will be recorded in wakefulness and sleep.
  Interventions: Behavioral: Prolonged wakefulness
- Sleep deprivation older men (Experimental): Older study participants will complete four nights in the sleep laboratory, whereas they will stay awake during one night. PET brain imaging will be conducted at the same circadian time on three consecutive afternoons (prior, during and after prolonged wakefulness). Additionally, validated tests of vigilance and cognitive performance will be administered and the brain waves will be recorded in wakefulness and sleep.
  Interventions: Behavioral: Prolonged wakefulness

INTERVENTIONS:
Behavioral: Prolonged wakefulness — 40 hours of prolonged wakefulness

SUMMARY:
A sleep deprivation protocol combined with state-of-the-art, simultaneous positron emission tomography and magnetic resonance spectroscopy imaging will be employed to investigate the effects of sleep deprivation and aging on hypothesized molecular markers of sleep need.

ELIGIBILITY:
Inclusion Criteria:

* healthy male individuals
* age: 20-35 or 60-70 years
* right-handed
* non-smokers
* moderate caffeine/alcohol consumption
* normal BMI

Exclusion Criteria:

* Sleep/circadian rhythms disturbances
* former brain injuries with loss of consciousness and brain anomalies
* drug intake/consumption
* medication intake
* cardiac pacemaker
* neurological disorders
* prior participation (during past 2 years) in radiological or nuclear experiment

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sleep-wake induced change in cerebral availability of mGluR5 (metabotropic glutamate receptors of subtype 5) | Change from baseline metabotropic glutamate receptors of subtype 5 availability after 33 hours of prolonged wakefulness and 8 hours of recovery sleep
  Positron emission tomography

SECONDARY OUTCOMES:
Sleep-wake induced change in glutamate concentration in prefrontal cortex and basal ganglia | Change from baseline glutamate concentration after 33 hours of prolonged wakefulness and 8 hours of recovery sleep
  Magnetic resonance spectroscopy
Sleep-wake induced change in potential molecular markers of sleep need | Change from baseline microRNA, fragile X mental retardation protein and brain-derived neurotrophic factor concentrations after 33 hours of prolonged wakefulness and 8 hours of recovery sleep
  microRNAs, fragile X mental retardation protein, and brain-derived neurotrophic factor concentrations in peripheral blood
Sleep-wake induced change in sleep electroencephalogram (EEG) | Change from all-night baseline sleep EEG in 8 hours of recovery sleep after 33 hours of prolonged wakefulness
  Spectral composition of the EEG during sleep
Sleep-wake induced change in waking electroencephalogram (EEG) | Change from baseline waking EEG during 33 hours of prolonged wakefulness and after 8 hours of recovery sleep
  Spectral composition of the EEG in wakefulness
Sleep-wake induced change in subjective state | Change from baseline sleepiness during 33 hours of prolonged wakefulness and after 8 hours of recovery sleep
  Subjective sleepiness as quantified with the Stanford Sleepiness Scale (range: 1 to 7)
Sleep-wake induced change in cognitive performance | Change from baseline cognitive performance during 33 hours of prolonged wakefulness and after 8 hours of recovery sleep
  Cognitive performance battery including tasks measuring sustained attention, executive functioning and working memory

CONTACTS AND LOCATIONS:
Overall Officials: Hanspeter Landolt, Prof, Principal Investigator — University of Zurich, Institute of Pharmacology and Toxicology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weigend S, Holst SC, Treyer V, O'Gorman Tuura RL, Meier J, Ametamey SM, Buck A, Landolt HP. Dynamic changes in cerebral and peripheral markers of glutamatergic signaling across the human sleep-wake cycle. Sleep. 2019 Oct 21;42(11):zsz161. doi: 10.1093/sleep/zsz161. PMID 31304973